CLINICAL TRIAL: NCT02144233
Title: Restoring Masticatory Function as Treatment for Chronic Pain: a Randomized Placebo-controlled Trial
Brief Title: Restoring Masticatory Function to Treat Chronic Pain
Acronym: MAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis showed benefice of one therapy over the other one.
Sponsor: Urbano Santana Penin, MD, DDS, PhD (Other)
Collaborators: University of Santiago de Compostela (Other)
Responsible Party: Sponsor-Investigator, Urbano Santana Penin, MD, DDS, PhD, Prof., University of Santiago de Compostela
Organization: University of Santiago de Compostela (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U1111-1134-0832; PI11/02507 (Other Grant/Funding Number: Ministry of Science and Innovation (Spain)); ISRCTN (Registry Identifier: 61654487)
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Results first posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Temporomandibular Joint Dysfunction Syndrome; Chronic Pain
Keywords: Pain; Temporomandibular joint disorders; Occlusal adjustment; Therapy; Randomized clinical trial; Mastication; Habitual chewing side; Handedness preference; Jaw asymmetry
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome; Chronic Pain; Pain; Temporomandibular Joint Disorders | interventions — Occlusal Adjustment

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Occlusal adjustment therapy (Experimental): Occlusal adjustment therapy consists of the elimination of premature tooth contacts during retruded jaw closure, and the reduction of the steeper lateral anterior guidance; the magnitude of this alteration will be estimated by the following equation: (right condylar path) × (left anterior guidance) = (left condylar path) × (right anterior guidance). A resin-composite, placed mainly in the canine tooth, can be used to increases the flatter lateral guidance on the habitual chewing side; overcorrection is expected to compensate for a masticatory preference on the opposite side to the handedness.
  Interventions: Procedure: Occlusal adjustment
- Placebo occlusal adjustment therapy (Placebo Comparator): Placebo occlusal adjustment will take place in a manner identical to the real adjustment. However, a specially fabricated inactive rotary instrument will be used, and no enamel will be removed.
  Interventions: Procedure: Placebo occlusal adjustment

INTERVENTIONS:
Procedure: Occlusal adjustment — The first step consists of the elimination of premature tooth contacts during retruded jaw closure.
  The second step included reduction of the steeper lateral anterior guidance; the magnitude of this alteration will be estimated by the following equation: (right condylar path) × (left anterior guidance) = (left condylar path) × (right anterior guidance)
  Other Names: Occlusal reshaping; Selective grinding of teeth; Restoring physiological jaw-closure; Restoring impaired chewing function
  Arms: Occlusal adjustment therapy
Procedure: Placebo occlusal adjustment — Placebo occlusal adjustment will take place in a manner identical to the real adjustment. However, a specially fabricated inactive rotary instrument will be used, and no enamel will be removed.
  Arms: Placebo occlusal adjustment therapy

SUMMARY:
The primary endpoint will be the average change in pain score from baseline to the three- and six-month assessments. Efficacy will be demonstrated by superior pain relief with the active treatment compared with the placebo.

DETAILED DESCRIPTION:
* The cause of temporomandibular joint (TMJ) disorders (TMD) remains unknown and therapy is usually empirical. Systematic reviews have concluded that currently there is no evidence that occlusal adjustment has any therapeutic or preventive effect on temporomandibular disorders. However, these reviews also indicate that evidence to the contrary has not been provided and that more research is needed to elucidate whether there is any benefit of occlusal adjustment treatment for TMD. The risk factors for chronic unilateral TMD include a steeper condylar path, flatter lateral anterior guidance, and habitual chewing on the affected side. Consequently, a new occlusal therapy is proposed to restore the physiological jaw closure and masticatory function.
* The primary end point of the trial is to assess the efficacy of the new occlusal therapy on the affected side TMD pain, and the maximum mouth opening. Efficacy is demonstrated by showing significantly superior pain relief and increasing maximum mouth opening (when it was limited) with the active treatment compared with placebo.

Phase III, single center, randomized, parallel-group, single-blind with blinded assessment, placebo-controlled clinical trial.

* A linear mixed model will be performed for comparisons of most variables and a logistic regression model will be used to measure the probability/risk of change on the chewing side between baseline and six months; in addition, McNemar's test may be used.
* Interim analysis plan and stopping rules. The study will employ an interim analysis plan with a single interim analysis after 70% of participants have completed the six-month follow-up visit. Using the Lan-DeMets version of the O'Brien-Fleming stopping rule, the critical value for statistical significance at the interim analysis (under intention-to-treat approach) will be +2.438, corresponding to a nominal two-sided P value of 0.0146.

Participants remaining with significant pain (and/or limited mouth opening) after the study will be invited to follow the conventional treatment, or to "complete" occlusal adjustment (rescue therapy): the full adjustment (if they were placebos), or a refining (if they received real therapy); the kind of received therapy will not be disclosed to participants. It based on the researchers' conviction, participants are encouraged to receive electively "complete" occlusal adjustment. All participants will be reevaluated between 3 to 6 months after study (12-Mo follow-up). Although no pain was reported at the 6-Mo follow-up, if pain returns, same approach will be carried out. Two sessions occlusal adjustment will be carried out and, if the pain remains, the patient will be treated following the Hospital approaches. The evolution of patients during post-MAP period, until writing of the manuscript, will be reported in the same manuscript, even if MAP result early stopped.

Additional patient's monitoring until next five years after treatment is expected.

ELIGIBILITY:
Inclusion Criteria:

* Completely dentate (except for the third molars; including if they were treated before enrollment by conventional or implant-supported fixed prosthesis allowing similar potential comfortable chewing on both sides)
* Normal Angle Class I occlusion
* Self-reported pain-intensity scores from 4 to 9 in a 0-10 visual analogue scale (VAS) or numerical pain rating scale (NRS).
* Chronic (over 6 months) joint and/or muscle pain, according to diagnostic criteria for temporomandibular disorders (DC/TMD), for which they had requested therapy

Exclusion Criteria:

* Psychosis
* Major depression
* Substance abuse
* Cognitive impairment
* Addiction to morphine or derivates
* Litigation or asking for disability/retirement compensation for chronic pain
* Dental care professionals
* Orthodontic therapy during the last 2 years
* Patients with any pain that is more severe, in the same location as, or cannot be clearly distinguished from TMD pain
* Individuals for whom minimally invasive occlusal adjustment could not achieve occlusal equilibration, including: Over 2 mm of difference between the maximal intercuspal position and the centric occlusion or over 4 mm of difference between upper and lower archs (or over 2mm on at less one side) measured: between the mesial fosses of first upper premolars with respect the buccal cusps of the first lower premolars; and/or between the mesiopalatal cusp of the first upper molars respect to the central (mesial) fossae of the first lower molar.
* Severe periodontal disease with grade 3 mobility

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Urbano Santana-Penin, Prof, Principal Investigator — University of Santiago de Compostela; Jose Lopez-Cedrun, Dr, Study Chair — University Hospital Complex of La Coruña; Maria J Mora, Prof, Study Director — University of Santiago de Compostela; Urbano Santana-Mora, Dr, Principal Investigator — University of Santiago de Compostela
Locations (2):
- Spain (2):
  - Universidad de Santiago de Compostela, Santiago de Compostela, A Coruña, Galicia
  - Complexo Hospitalario Universitario A Coruña, A Coruña, A Coruña. Galicia

IPD SHARING:
Plan to Share IPD: Yes
A closed, certificate, database called OpenClinica allows access to members of the Data and Safety Monitoring Board.
  We expect to publish raw data in Sci Data. Figures from participant's mouth could be posted in a repository. The protocol will be attached as a supplementary appendix to the main manuscript
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The raw data of each participant, unidentifiable, will be accessible within 6 months after the publication of the manuscript and will be accessible for at least one year.
Access Criteria: Free access

REFERENCES:
- [Background] Santana-Mora U, Lopez-Cedrun J, Mora MJ, Otero XL, Santana-Penin U. Temporomandibular disorders: the habitual chewing side syndrome. PLoS One. 2013 Apr 8;8(4):e59980. doi: 10.1371/journal.pone.0059980. Print 2013. PMID 23593156

RESULTS

PARTICIPANT FLOW:
Groups:
- Occlusal Adjustmen Therapy: Occlusal adjustment therapy consists of the elimination of premature tooth contacts during retruded jaw closure, and the reduction of the steeper lateral anterior guidance; the magnitude of this alteration will be estimated by the following equation: (right condylar path) × (left anterior guidance) = (left condylar path) × (right anterior guidance). A resin-composite, placed mainly in the canine tooth, can be used to increases the flatter lateral guidance on the habitual chewing side; overcorrection is expected to compensate for a masticatory preference on the opposite side to the handedness.
  Occlusal adjustment: The first step consists of the elimination of premature tooth contacts during retruded jaw closure.
  The second step included reduction of the steeper lateral anterior guidance; the magnitude of this alteration will be estimated by the following equation: (right condylar path) × (left anterior guidance) = (left condylar path) × (right anterior guidance)
Period: Overall Study
Arm/Group | Occlusal Adjustmen Therapy | Placebo Occlusal Adjustment Therapy
Started | 39 | 38
Completed | 39 (The last participant was assessed at month 3 due to early study stop) | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Occlusal Adjustmen Therapy: Occlusal adjustment therapy consists of the elimination of premature tooth contacts during retruded jaw closure, and the reduction of the steeper lateral anterior guidance; the magnitude of this alteration will be estimated by the following equation: (right condylar path) × (left anterior guidance) = (left condylar path) × (right anterior guidance). A resin-composite, placed mainly in the canine tooth, can be used to increases the flatter lateral guidance angle on the habitual chewing side; overcorrection is expected to compensate for a masticatory preference on the opposite side to the handedness.
  Occlusal adjustment: The first step consists of the elimination of premature tooth contacts during retruded jaw closure.
  The second step included reduction of the steeper lateral anterior guidance; the magnitude of this alteration will be estimated by the following equation: (right condylar path) × (left anterior guidance) = (left condylar path) × (right anterior guidance)
- Total: Total of all reporting groups
Arm/Group | Occlusal Adjustmen Therapy | Placebo Occlusal Adjustment Therapy | Total
Number analyzed (Participants) | 39 | 38 | 77
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 29 [22 to 38] | 30 [25 to 40] | 30 [24 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 35 | 72
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 38 | 36 | 74
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Self-reported jaw-pain intensity [Median (Inter-Quartile Range); unit: units on a 0-10 scale] — Self-reported pain-intensity on the affected side measured by the Visual Analogue Scale (VAS) and/or Numerical Pain Rating Scale (NRS). We will work with a 0-10 scale, with 0 indicating no-pain and 10 the worst possible pain.
  units on a 0-10 scale | 7 [5 to 8] | 7 [6 to 7] | 7 [6 to 7]

OUTCOME MEASURES:

1. Primary Outcome: Jaw-pain-Intensity (Affected Side)
Description: Self-reported affected-side pain-intensity across the trial in a 0-10 visual analogue scale (VAS) (0=no pain, 10=worst possible pain). Higher values represent a worse outcome.
Time Frame: Baseline and 6-months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Occlusal Adjustmen Therapy: Occlusal adjustment therapy consists of the elimination of premature tooth contacts during retruded jaw closure, and the reduction of the steeper lateral anterior guidance; the magnitude of this alteration will be estimated by the following equation: (right condylar path) × (left anterior guidance) = (left condylar path) × (right anterior guidance). A resin-composite, placed mainly in the canine tooth, can be used to increases the flatter LG on the habitual chewing side; overcorrection is expected to compensate for a masticatory preference on the opposite side to the handedness.
  Occlusal adjustment: The first step consists of the elimination of premature tooth contacts during retruded jaw closure.
  The second step included reduction of the steeper lateral anterior guidance; the magnitude of this alteration will be estimated by the following equation: (right condylar path) × (left anterior guidance) = (left condylar path) × (right anterior guidance)
Arm/Group | Occlusal Adjustmen Therapy | Placebo Occlusal Adjustment Therapy
Number analyzed (Participants) | 39 | 38
units on a scale
  baseline | 7 [5 to 8] | 7 [6 to 7]
  6-Months | 2 [0 to 3] | 3.5 [1 to 6]

2. Secondary Outcome: Chewing Side
Description: A consistent chewing side was considered if at lees 5 out of 7 almonds (or at lees 7 of 10 cycles of chewing gum), the participant report to use same side, and same side was used during kinesiography recordings of spontaneous chewing. Any other results lead to alternate chewing allocation.
Time Frame: Baseline and 6-months
Measure: Count of Participants; unit: Participants
Arm/Group | Occlusal Adjustmen Therapy | Placebo Occlusal Adjustment Therapy
Number analyzed (Participants) | 39 | 38
Participants
  baseline: Right | 16 | 14
  baseline: Alternate | 8 | 13
  baseline: Left | 15 | 11
  6-Months: Right | 6 | 6
  6-Months: Alternate | 25 | 27
  6-Months: Left | 8 | 5

3. Secondary Outcome: Change in Global Severity Index Scores (Symptom Checklist-90-Revised (SCL-90-R))
Description: Mean change in Global Severity Index scores from a self-administered Spanish validated questionaire SCL-90-R. Higher values represent a worse outcome. Range (0-4).
Time Frame: Baseline, 6-Months
Population: Some self administered questionnaire was not adequately covered by the patient.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Occlusal Adjustmen Therapy | Placebo Occlusal Adjustment Therapy
Number analyzed (Participants) | 39 | 38
score on a scale
  baseline: number analyzed (Participants) | 39 | 37
  baseline | 0.89 (0.57) | 0.81 (0.51)
  6-Months: number analyzed (Participants) | 37 | 34
  6-Months | 0.52 (0.5) | 0.5 (0.49)
Statistical Analysis 1: Comparison: Occlusal Adjustmen Therapy vs Placebo Occlusal Adjustment Therapy; Test type: Superiority; p = 0.54, Mixed Models Analysis

4. Secondary Outcome: Maximum Unassisted Jaw Opening
Description: Vertical jaw-opening (incisal level) measured using a ruler. Higher values represent a better outcome.
Time Frame: Baseline, 3- and 6-Months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Occlusal Adjustmen Therapy | Placebo Occlusal Adjustment Therapy
Number analyzed (Participants) | 39 | 38
mm
  baseline | 41.5 (8.4) | 43.9 (7.8)
  3-Months | 45.66 (7.9) | 46.73 (7.7)
  6-Months | 47.7 (8.4) | 46.4 (7.7)

5. Other Pre Specified Outcome: Headache-intensity
Description: Headache intensity in recent months (If any) in a 0-10 numerical pain rating scale with 0=no pain and 10= worst possible pain.
Time Frame: Baseline 3- and 6-Months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Occlusal Adjustmen Therapy | Placebo Occlusal Adjustment Therapy
Number analyzed (Participants) | 39 | 38
score on a scale
  baseline | 7 [5 to 8] | 5.75 [1 to 7.63]
  3-Months | 4 [1.5 to 6] | 3 [0.5 to 6]
  6-Months | 4 [0 to 5] | 3 [0 to 7]

6. Other Pre Specified Outcome: Number of Participants With Neuropathic Pain
Description: Neuropathic pain Questionnaire (DN4). Over 4 scores indicates neuropathic facial pain.
Time Frame: Baseline, 6-Months
Population: Data from 1 placebo group participant at 6-months not available
Measure: Count of Participants; unit: Participants
Arm/Group | Occlusal Adjustmen Therapy | Placebo Occlusal Adjustment Therapy
Number analyzed (Participants) | 39 | 37
Participants
  baseline: neuropathic pain | 13 | 12
  baseline: without neuropathic symptoms | 26 | 25
  at month 6: neuropathic pain | 3 | 4
  at month 6: without neuropathic symptoms | 36 | 33

7. Other Pre Specified Outcome: Handedness Preference
Description: Handedness preference assessed using Edinburg inventory:
  Left Right
  1. Writing
  2. Drawing
  3. Throwing
  4. Scissors
  5. Toothbrush
  6. Knife (without fork)
  7. Spoon
  8. Broom (upper hand)
  9. Striking Match (match)
  10. Opening box (lid) I Which foot do you prefer to kick with? II Which eye do you use when using only one?
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Occlusal Adjustmen Therapy | Placebo Occlusal Adjustment Therapy
Number analyzed (Participants) | 39 | 38
Participants
  right | 29 | 31
  left | 10 | 7

8. Other Pre Specified Outcome: Lateral Guidance Angles (LG)
Description: The angle between the tangent of the LG tracings and the horizontal Frankfort line, starting from the midsagittal point up 2 mm: using a calibrated Model K7 diagnostic system. Both sides recordings of each patient were measured and considered individually. The mean of both sides of each patient was not used.
Time Frame: Baseline
Population: Note that both sides of each participant was assessed. Recordings from one participant in each group are unavailable.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: LG
Arm/Group | Occlusal Adjustmen Therapy | Placebo Occlusal Adjustment Therapy
Number analyzed (Participants) | 38 | 37
Number analyzed (LG) | 76 | 74
degrees | 42 (10.3) | 40.6 (11.8)

9. Other Pre Specified Outcome: Condylar Path Angles
Description: Parasagittal plane condylar path tracings in relation to the Frankfort Horizontal Plane following the Gysi extraoral method.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Occlusal Adjustmen Therapy | Placebo Occlusal Adjustment Therapy
Number analyzed (Participants) | 39 | 38
degrees
  right joint | 50.5 (10.7) | 47.3 (8.1)
  left joint | 50.1 (10.5) | 49.3 (8.6)

10. Other Pre Specified Outcome: Adverse Events
Description: Unexpected Adverse Events (NIH, 2009).
Time Frame: After therapy, 1-Month, 3-Months, 6-Months
Measure: Count of Participants; unit: Participants
Arm/Group | Occlusal Adjustmen Therapy | Placebo Occlusal Adjustment Therapy
Number analyzed (Participants) | 39 | 38
Participants | 0 | 0

11. Other Pre Specified Outcome: Jaw Asymmetry
Description: Over 1 mm of interincisal midline deviation and inter-arches Angle Classification of the lateral sectors (canines and first molars); it will be assessed during maximal intercuspal position and during jaw retruded contact position
Time Frame: Baseline
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Participant's Awareness With Trial Group Assignment
Description: Physicians and patients are quizzed at the end of the study to determine whether or not they have guessed the therapy involved
Time Frame: Six months
Measure: Count of Participants; unit: Participants
Arm/Group | Occlusal Adjustmen Therapy | Placebo Occlusal Adjustment Therapy
Number analyzed (Participants) | 39 | 38
Participants
  real therapy | 26 | 21
  I don't' know | 12 | 14
  placebo therapy | 1 | 3

13. Other Pre Specified Outcome: Credibility (of Participants)
Description: Confidence of participants in the goodness of treatment.
  These items were simplified here to the following single question:
  How confident would you be that this treatment would be successful in eliminating your pain and/or limited mouth opening? 0-10 numerical rating scale, with 0=nothing to 10= totally.
Time Frame: Baseline, 6-Months
Population: Data from one participant from each group was lost from baseline, and 2 from the Occlusal adjustment group and 5 from the placebo group at 6-months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Occlusal Adjustmen Therapy | Placebo Occlusal Adjustment Therapy
Number analyzed (Participants) | 37 | 33
units on a scale
  baseline | 8 (1.8) | 8.3 (1.3)
  6-Months | 8 (1.9) | 7.6 (2.6)

14. Other Pre Specified Outcome: Sociodemography
Description: Level of education
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Occlusal Adjustmen Therapy | Placebo Occlusal Adjustment Therapy
Number analyzed (Participants) | 39 | 38
Participants
  Higher | 21 | 26
  Secondary | 12 | 9
  No qualifications | 6 | 3

15. Other Pre Specified Outcome: Patient Impression (Improvement)
Description: Patient impression outcome will be reported as Improved Vs. no change.
Time Frame: 6-Months
Population: Data from two participants in placebo group that underwent randomization were not available.
Measure: Count of Participants; unit: Participants
Arm/Group | Occlusal Adjustmen Therapy | Placebo Occlusal Adjustment Therapy
Number analyzed (Participants) | 39 | 36
Participants
  Improved | 37 | 25
  No change | 2 | 11

16. Other Pre Specified Outcome: Pain Interference on Daily Activity
Description: In the past 6 months, how much has facial pain interfered with your daily activities rated on a 0-10 scale where 0 is "no interference" and 10 is "unable to carry on any activities"? 0-10 VAS/NRS (0=No interference to 10=Unable to carry on any activities). N.B. Only one item was choose to simplify.
Time Frame: Baseline; 6-Months
Population: Data from two occlusal adjustment and six placebo group participants were not available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Occlusal Adjustmen Therapy | Placebo Occlusal Adjustment Therapy
Number analyzed (Participants) | 37 | 32
units on a scale
  baseline | 5.2 (2.6) | 4.5 (2.9)
  6-Months | 3.1 (2.6) | 2 (3.2)

17. Other Pre Specified Outcome: Pain-dimensions
Description: McGill Pain questionnaire
Time Frame: Baseline, 6-Months
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Temporomandibular Disorders Related Impairment
Description: Mandibular Function Impairment Questionnaire (MFIQ)
Time Frame: Baseline, 6-Mo
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Circulating Biomarkers
Description: Blood levels of Circulating Biomarkers
Time Frame: Baseline, 6-Months
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Periodontal Disease (if Indicated)
Description: Radiographic defect, Probing depth, Clinical attachment level, Tooth mobility Tooth mobility
Time Frame: Baseline, 6-Months
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Occlusal Forces/Pressure
Description: Dental or occlusal forces measured using fuji-film method.
Time Frame: Baseline; 6-Months
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Maximum Comfortable (Without Pain) Jaw Opening
Description: Vertical jaw-opening (incisal level) measured using a ruler.
Time Frame: Baseline, immediate after therapy, 3- and 6-Months
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Patient's Perception of Reduced Movement
Description: Subjective patient's perception of reduced jaw-opening; how many fingers can put between your incisors?. Higher values represent a better outcome.
Time Frame: Baseline, 6-Months
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Protrusive Motion
Description: Magnitude (mm) of protrusive jaw-movement (incisal level) and lateral shift (quantitative, mm; and/or qualitative, left/right), using kinesiography recordings. Higher values represent a better outcome.
Time Frame: Baseline, 6-Months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Description: The dental hypersensitivity period (referred to as discomfort to the chewing foods crisp) lasted between 1 and 3 months.
Arm/Group | Occlusal Adjustmen Therapy | Placebo Occlusal Adjustment Therapy
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/38
Other Adverse Events (participants affected / at risk) | 3/39 | 0/38
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Occlusal Adjustmen Therapy (N=39) | Placebo Occlusal Adjustment Therapy (N=38)
Dental hypersensitivity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) — Dental hypersensitivity, treated using topic fluorides

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT02144233/Prot_SAP_000.pdf